CLINICAL TRIAL: NCT02563145
Title: Real-time fMRI for the Treatment of Aggressive Behavior in Adolescents (Part of EU-MATRICS: Multidisciplinary Approaches to Translational Research)
Brief Title: Real-time fMRI for the Treatment of Aggressive Behavior in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU Health-F2-2013-603016
Record Dates: First submitted 2015-09-28; First posted 2015-09-29 (Estimated); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Aggression; Conduct Disorder
Keywords: Real-time fMRI feedback
MeSH Terms: conditions — Aggression; Conduct Disorder | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Real-time fMRI feedback (Experimental): After a pre-training assessment at baseline, subjects will be randomized to either treatment arm or treatment as usual. Subjects in the experimental condition will receive 10 sessions of real-time fMRI feedback of insula- or amygdala activation (dependent on activation patterns during pre-testing), 1 session/week. Each session will last about 1 1/2 hours.
  After training completion (10 weeks after the beginning of the treatment phase), subjects will undergo post-treatment assessment and follow up (6 months after the end of the training phase).
  Interventions: Behavioral: Real-time fMRI feedback
- Treatment as usual (Active Comparator): After a pre-training assessment at baseline, subjects will be randomized to either treatment arm or treatment as usual. Subjects in the comparator TAU arm will receive several sessions of psychoeducation and counseling with their parents/caregivers or group training over 10 weeks.
  Within the sessions, investigators will focus on psychoeducational issues and provide general counseling for the families. After 10 weeks, subjects will undergo post-treatment assessment and follow up (6 months after the end of the treatment phase).
  Interventions: Behavioral: Treatment as usual
- Typically developing (TD) control group (No Intervention): Healthy typically developing subjects will only participate in pre-training assessment to allow for comparison.

INTERVENTIONS:
Behavioral: Real-time fMRI feedback — feedback about activation patterns in brain regions related with instrumental aggression
  Arms: Real-time fMRI feedback
Behavioral: Treatment as usual — Psychoeducation, general counselling
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to determine whether real-time fMRI feedback is effective in the treatment of aggressive behavior problems in adolescents with high callous unemotional traits when compared to treatment as usual.

DETAILED DESCRIPTION:
In this study, which is part of the European research project MATRICS (Multidisciplinary Approaches to Translational Research), the investigators focus on testing an innovative, non-pharmacological therapeutic approach for adolescents with a specific, difficult to treat subtype of aggressive behavior problems. Participants will be trained to acquire control over their own physiological parameters, in case of this study the activation of certain brain areas. While trying to control these parameters, participants get direct continuous feedback about their physiological state and its changes, and are rewarded for successful manipulation. Biofeedback methods are currently used to treat patients with a variety of psychiatric disorders such as attention-deficit/hyperactivity disorder (ADHD).

Here, real-time functional magnetic resonance imaging (rt-fMRI) feedback will be used, where participants will get feedback about activation levels and patterns from brain regions associated with emotion processing (amygdala/insula) in almost real time while lying in a magnetic resonance tomograph scanner.

Investigators will focus on the following questions concerning the effectiveness of this treatment approach:

1. Can participants gain increasing control over the activation of defined brain regions through real-time fMRI training?
2. Which short- and longer term consequences can be expected from improved self control over brain activation upon aggressive and antisocial behavior problems?

Before the training, all participants will undergo an extensive pre-treatment assessment as part of the characterization and subtyping of aggression within the large multicenter subtyping studies (EU-Aggressotype and EU-MATRICS). The assessment includes clinical and psychometric measures, neuropsychological testing, fMRI (3 active tasks + resting state), MRS (anterior cingulate cortex (ACC) and insula) and diffusion tensor imaging (DTI) as well as biosampling (blood/saliva for genetics/epigenetics/hormones). Comparison with a typically developing (TD) control group receiving no intervention will allow to interpret changes in terms of normalization or compensation.

After completion of this pretest, subjects meeting the inclusion criteria for the rt-fMRI treatment study will be randomly assigned to two different treatment arms, either to the experimental fMRI real-time feedback condition or to the comparator condition with treatment as usual (TAU) lasting 10 weeks. Subjects assigned to the experimental condition will receive 10 sessions (1/week) of real-time fMRI feedback of amygdala and/or insula activation (based on activation patterns during pre-training assessment). Each training will last about 1 1/2 hours and consist of 3 experimental blocks, including feedback- and transfer trials. Video clips of emotional and aggressive interpersonal interactions will partly be used to enrich feedback conditions with naturalistic, virtual reality type displays. Heart rate and electrodermal activity will be recorded simultaneously during the sessions. Subjects in the comparator TAU arm will receive several sessions of psychoeducation and counseling with their parents/caregivers or group training over the 10 weeks.

After completion of either the training or the TAU, subjects will undergo post-treatment assessment, repeating the teachers and parents reports on behavioral measures, as well as the neuropsychological testing, fMRI and MRS. A follow-up assessment will take place 6 months after the end of the treatment phase and will comprise only parents and teachers reports on behavioral measures.

ELIGIBILITY:
Inclusion Criteria (interventional group):

* ODD/CD diagnosis based on the DSM-5 criteria
* aggression in the clinical range, T > 70 on the aggression or delinquency subscale of the Teacher Report Form (TRF), Youth Self Report (YSR) or Child Behaviour Checklist (CBCL)
* preferably medication-naive, otherwise medication should be stable for at least 2 months

Inclusion Criteria (typically developing (TD) group):

* no diagnosis based on the DSM-5 criteria
* aggression below the clinical range, T < 70 on the aggression or delinquency subscale of the Teacher Report Form (TRF), Youth Self Report (YSR) or Child Behaviour Checklist (CBCL)

Exclusion Criteria (both groups):

* IQ<80
* a primary DSM-5 diagnosis of psychosis, bipolar disorder, depression or anxiety
* contra-indications for MRI scanning, e.g. presence of metal parts in the body
* epilepsy

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2015-10; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Changes in aggressive behavior from baseline at 10 weeks and 6 months as assessed by the Modified Overt Aggression Scale (MOAS) | Baseline, post treatment assessment (10 weeks after beginning of the treatment phase) and follow up (6 months after end of the treatment)
  Parents or caregivers report on type and intensity of aggressive behavior over the last weeks (questionnaire)

SECONDARY OUTCOMES:
Changes in brain activation from baseline at 10 weeks after the beginning of the treatment phase as assessed by fMRI | Baseline and post treatment assessment (10 weeks after the beginning of the treatment phase)
  At baseline and at the end of the treatment phase, patients will perform 3 functional tasks in the fMRI. The tasks used are: Stop-Signal Task, Emotional Faces task, Passive Avoidance task.
Changes in composition of neurotransmitter systems from baseline at 10 weeks after the beginning of the treatment phase as assessed by MRS | Baseline and post treatment assessment (10 weeks after the beginning of the treatment phase)
  At baseline and at the end of the treatment phase, patients will undergo magnetic resonance spectroscopy (MRS) of two brain areas implicated in inhibitory control (ACC and insula)
Changes in aggressive behavior from baseline at 10 weeks and at 6 months as reported by teachers through the aggressive behavior subscale of the TRF (Teachers Report Form) | Baseline, post treatment assessment (10 weeks after beginning of the treatment phase) and follow up (6 months after end of the treatment)
  At baseline, after the end of the treatment phase (10 weeks) and at follow up (6 months), teachers will be asked to complete the TRF, which is a questionnaire focusing on general psychopathology ( and allows to differentiate between several subsets of symptoms, amongst others those indicating externalizing and aggressive behavior)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Brandeis, PhD, Principal Investigator — Department of Child and Adolescent Psychiatry and Psychotherapy, CIMH Medical Faculty Mannheim/ Heidelberg University, Mannheim, Germany; Tobias Banaschewski, MD, PhD, Principal Investigator — Department of Child and Adolescent Psychiatry and Psychotherapy, CIMH Medical Faculty Mannheim/ Heidelberg University, Mannheim, Germany
Locations (1):
- Department of Child and Adolescent Psychiatry and Psychotherapy, CIMH Medical Faculty Mannheim/ Heidelberg University, Mannheim, Germany, Mannheim, Germany